CLINICAL TRIAL: NCT06711913
Title: Effects of Intravenous Dexmedetomidine on Shivering After Cesarean Delivery Under Neuraxial Anesthesia - A Randomized Control Trial
Brief Title: Role of Intravenous Dexmedetomidine in Reducing Shivering After Shivering Cesarean Section Due to Spinal Anesthesia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Liaquat National Hospital & Medical College (Other)
Responsible Party: Principal Investigator, Ghulam Fatima, Principal Investigator, Liaquat National Hospital & Medical College
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Liaquat National Hospital 1234; Dr ghulam fatima (Other: liaquat national hospital)
Record Dates: First submitted 2024-11-21; First posted 2024-12-02 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Shivering
Keywords: shivering, dexmedetomidine, neuraxial anesthesia
MeSH Terms: interventions — Dexmedetomidine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Active Comparator): Received intravenous dexmedetomidine
  Interventions: Drug: Dexmedetomidine
- Control group (Placebo Comparator): control group receive normal saline
  Interventions: Other: Normal Saline (Placebo)

INTERVENTIONS:
Drug: Dexmedetomidine — intravenous dexmedetomidine given in form of 100ml infusion over 10 minutes
  Arms: Intervention group
Other: Normal Saline (Placebo) — control group receive normal saline as placebo
  Arms: Control group

SUMMARY:
"After spinal anesthesia, some patients may experience shivering, which can be uncomfortable and even lead to complications. Dexmedetomidine is a medication that can help prevent or reduce this shivering.

Dexmedetomidine helps to:

1. Reduces shivering and discomfort.
2. Improves patient comfort and satisfaction.
3. Regulates body temperature.
4. Safe and effective.

DETAILED DESCRIPTION:
Post-spinal shivering is a common complication that occurs in 40-65% of patients undergoing spinal anesthesia. It is characterized by involuntary, rhythmic muscle contractions that can lead to discomfort, anxiety, and increased oxygen consumption.

The exact mechanisms underlying post-spinal shivering are not fully understood, but several factors contribute to its development:

1. *Hypothermia*: Spinal anesthesia can cause a decrease in core body temperature, leading to shivering.
2. *Sympathetic blockade*: Spinal anesthesia blocks sympathetic nerve fibers, causing vasodilation and decreased blood flow to the extremities.
3. *Increased oxygen consumption*: Shivering increases oxygen consumption, which can be detrimental in patients with pre-existing cardiovascular or respiratory disease.

*Effects of Dexmedetomidine on Post-Spinal Shivering*

Dexmedetomidine, an alpha-2 adrenergic agonist, has been shown to effectively reduce post-spinal shivering. Its effects include:

1. *Decreased shivering intensity*: Dexmedetomidine reduces the severity of shivering, making patients more comfortable.
2. *Increased core body temperature*: Dexmedetomidine helps to maintain core body temperature, reducing the likelihood of hypothermia-induced shivering.
3. *Reduced oxygen consumption*: By decreasing shivering, dexmedetomidine reduces oxygen consumption, which is beneficial for patients with cardiovascular or respiratory disease.
4. *Improved patient comfort*: Dexmedetomidine's sedative and anxiolytic effects contribute to improved patient comfort and satisfaction.
5. *Reduced need for other anti-shivering interventions*: Dexmedetomidine's effectiveness in reducing post-spinal shivering may reduce the need for other interventions, such as meperidine, clonidine, or forced-air warming.

Dexmedetomidine's anti-shivering effects are thought to be mediated by its actions on the following mechanisms:

1. *Alpha-2 adrenergic receptors*: Dexmedetomidine activates alpha-2 adrenergic receptors, which decreases sympathetic outflow and reduces shivering.
2. *Hypothalamic thermoregulation*: Dexmedetomidine may affect the hypothalamus, the body's thermoregulatory center, to reduce shivering and maintain core body temperature.
3. *Spinal cord mechanisms*: Dexmedetomidine may also act on the spinal cord to reduce shivering, possibly by inhibiting the release of excitatory neurotransmitters.

ELIGIBILITY:
Inclusion Criteria:

* Elective Cesarean section
* Age limit 18 to 35 years
* ASA II

Exclusion Criteria:

* Emergency cesarean delivery
* hypersensitive to dexmedetomidine
* Pateint with hear, renal, or hepatic diseases requiring follow up
* Pre-eclemptic pateint
* Patient with GA
* Combined spinal epidural anesthesia

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 60 (Actual)
Dates: Start 2023-12-21 (Actual); Primary Completion 2024-06-15 (Actual); Study Completion 2024-06-21 (Actual)

PRIMARY OUTCOMES:
Shivering | 3 minutes following infusion
  Crossley and Mahajan grading of intraoperative shivering Grade 0: no shivering grade 1:no visible muscle activity but piloerection, peripheral vasoconstriction, or both present grade 2: muscular activity in one muscle group grade 3: muscle activity in one than more muscle group

CONTACTS AND LOCATIONS:
Overall Officials: Ghulam Fatima kharl, Principal Investigator — Liaquat national hospital and medical college
Locations (1):
- Liaquat National Hospital and Medical College, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No
Reasons of why individual participant data (IPD) may not be shared:
  1. *Patient confidentiality*: Sharing IPD could compromise patient confidentiality
  2. *Informed consent*: Participants may not have provided informed consent for their data to be shared, which could raise ethical concerns.
  3. *Data storage and security*: Sharing IPD requires ensuring the security and integrity of the data, which can be a significant technical challenge.

REFERENCES:
- See also: Kumar S, Choudhury B, Varikasuvu SR, Singh H, Kumar S, Lahon J, et al. A Systematic Review and Meta-analysis of Efficacy and Safety of Dexmedetomidine Combined With Intrathecal Bupivacaine Compared to Placebo. Cureus. 2022;14(12):e32425. — https://doi.org/10.7759/cureus.32425